CLINICAL TRIAL: NCT00497328
Title: An Open Labelled Randomized Multi-center Study of COmbined N-acetylcysteine and Bicarbonate in PCI To Reduce Incidence of Contrast Induced Nephropathy
Brief Title: COmbined N-acetylcysteine and Bicarbonate in PCI To Reduce Adverse Side Effect of contrasT
Acronym: CONTRAST
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SQCIN01
Record Dates: First submitted 2007-07-04; First posted 2007-07-06 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Contrast Induced Nephropathy
Keywords: contrast induced nephropathy
MeSH Terms: interventions — Acetylcysteine; Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- N-acetylcysteine Group (NAC) (Other): N-acetylcysteine Group (NAC)
  Intravenous infusion 154mEq/L of sodium chloride (0.9% normal saline) at a rate of 1mL/kg/hour from 12 hours before till 6 hours after cardiac catheterization Oral NAC 1200mg dissolve in 250ml of water twice a day the day before to the day after the procedure (total 6 doses)
  Interventions: Drug: N-acetylcysteine
- Sodium Bicarbonate Group (SOB) (Other): Sodium Bicarbonate Group (SOB)
  Intravenous infusion154meq/L sodium bicarbonate in 5% dextrose in water at a rate of 3 mL/kg/hour for 1 hour immediately before radiocontrast injection. For patients weighing more than 110 kg, the initial fluid bolus and drip will be limited to those doses administered to a patient weighing 110 kg.
  Intravenous infusion154meq/L sodium bicarbonate in 5% dextrose in water at a rate of 1 mL/kg/hour during the contrast exposure and for 6 hours after the procedure
  Interventions: Drug: Sodium Bicarbonate
- Combination Group (COM: NAC and SOB) (Other): Combination Group (COM: NAC and SOB)
  Intravenous infusion of 154 meq/l sodium bicarbonate at a rate of 3ml/kg/hour for 1 hour before cardiac catheterization and 1 ml/kg/hour till 6 hours after procedure Oral NAC 1200mg dissolve in 250ml of water twice a day the day before to the day after the procedure (total 6 doses). All patients will be monitored regularly for pulmonary congestion and hemodynamics compromise hourly after PCI for 6 hours and every 4 hour thereafter for 24 hours.
  Interventions: Drug: N-acetylcysteine; Drug: Sodium Bicarbonate

INTERVENTIONS:
Drug: N-acetylcysteine
  Arms: Combination Group (COM: NAC and SOB); N-acetylcysteine Group (NAC)
Drug: Sodium Bicarbonate
  Arms: Combination Group (COM: NAC and SOB); Sodium Bicarbonate Group (SOB)

SUMMARY:
This is a randomised controlled trial to investigate the efficacy of preventive regimen of hydration with high dose oral N-acetylcysteine and intravenous sodium bicarbonate pretreatment in patients with stable advanced renal insufficiency (CKD stage 3 and 4:GFR 15-60ml/min/1.73m2 calculated by Modification of Diet in Renal Disease Study equation (MDRD formula)) undergoing elective percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
OBJECTIVES

Primary Objective To investigate whether combination therapy of high dose oral N-acetylcysteine NAC) and intravenous (IV) sodium bicarbonate can further reduce incidence of contrast induced nephropathy (CIN) in patients with baseline renal impairment undergoing elective percutaneous coronary intervention (PCI).

Secondary Objective

* To compare the effectiveness in prevention of CIN in either NAC or sodium bicarbonate arm of therapy.
* Maximum change in serum creatinine level within 30 days
* Difference in hospital stay between groups
* Need for hemodialysis within 30 days
* 30 day mortality
* Maximum change in GFR within 30 days
* Peak creatinine level within 48 hours and 30 days

TRIAL DESIGN Trial Design: Randomized, open label, active controlled, multi-center, efficacy study Trial Population: 630 Recruitment duration: 18 months

Trial Sites:

* National University Hospital (Singapore)
* Sarawak General Hospital (Malaysia)
* Institue Jantung Negara (Malaysia)
* Nanjing First Hospital (China)
* Guangdong Provincial Cardiovascular Institute (China) All patients with baseline creatinine clearance between 15 to 60 mL/min who undergo cardiac catheterization either electively or following acute coronary syndromes will be approached to participate in this study. After the written informed consent is signed, the patient will be screened for eligibility criteira. Only the eligible patients will be randomly assigned to one of three groups in 1:1:1 ratio.
* NAC: Infusion of sodium chloride and oral NAC
* SOB: Infusion of sodium bicarbonate
* COM: Infusion of sodium bicarbonate and oral NAC

Inclusion Criteria

* Age > 21 year
* Glomerular Filtration Rate (GFR) 15-60ml/min calculated by MDRD formula
* Scheduled to undergo elective PCI
* Able to receive 12 hours of pre-hydration
* Written informed consent

Exclusion Criteria:

* GFR less than 15ml/min or patients diagnosed with end stage renal failure
* Increase in serum creatinine levels of > 0.5mg/dl or 44umol/l in the previous 24 hours
* Preexisting dialysis
* Pulmonary edema or moderate to severe congestive heart failure (New York Heart Association [NYHA] III-IV)
* Patient unable to withstand the fluid load and hemodynamics compromise
* Uncontrolled hypertension (untreated systolic blood pressure > 160 mmHg, or diastolic blood pressure > 100mmHg.)
* Emergency cardiac catheterization (i.e. patient presenting with ST segment elevation myocardial infarction undergoing primary angioplasty)
* Recent exposure to radiographic contrast (within two days of the study).
* Allergic to radio-contrast
* Administration of sodium bicarbonate solution or NAC within 48 hours before the PCI.
* Patient unable to give consent
* Clinically vulnerable condition requiring continuous fluid therapy e.g. severe sepsis
* Use of NSAID, aminoglycocide, cyclosporin, cysplatin within 48 hours prior to PCI and throughout the study duration TREATMENT SCHEDULE

Treatment Groups

After randomisation, the patient will receive one of the following treatments:

N-acetylcysteine Group (NAC)

* Intravenous infusion 154mEq/L of sodium chloride (0.9% normal saline) at a rate of 1mL/kg/hour from 12 hours before till 6 hours after cardiac catheterization
* Oral NAC 1200mg dissolve in 250ml of water twice a day the day before to the day after the procedure (total 6 doses)

Sodium Bicarbonate Group (SOB)

* Intravenous infusion154meq/L sodium bicarbonate in 5% dextrose in water at a rate of 3 mL/kg/hour for 1 hour immediately before radiocontrast injection. For patients weighing more than 110 kg, the initial fluid bolus and drip will be limited to those doses administered to a patient weighing 110 kg.
* Intravenous infusion154meq/L sodium bicarbonate in 5% dextrose in water at a rate of 1 mL/kg/hour during the contrast exposure and for 6 hours after the procedure

Combination Group (COM: NAC and SOB)

* Intravenous infusion of 154 meq/l sodium bicarbonate at a rate of 3ml/kg/hour for 1 hour before cardiac catheterization and 1 ml/kg/hour till 6 hours after procedure
* Oral NAC 1200mg dissolve in 250ml of water twice a day the day before to the day after the procedure (total 6 doses). All patients will be monitored regularly for pulmonary congestion and hemodynamics compromise hourly after PCI for 6 hours and every 4 hour thereafter for 24 hours.

Trial Participation

Eligible subject will be enrolled in the study for 30 days. Assessments will be done on Day 1,2 and 3 (48 hours after PCI) and an end of study visit at Day 30.

Contrast used should be non-ionic low osmolality type (such as iohexol, iopamidol, ioversol,iopromide).

If the Day 3 serum creatinine level is increased to >25% above the baseline level (i.e.development of CIN), patient will continune to be monitored up to a week at the discretion of the investigator until serum creatinine level improved or CIN resolved.

Treatment Modification

All therapies will be discontinued should adverse-effects such as cardiac failure or pulmonary congestion develop, although these are anticipated to be at low event occurrence rate.

CONCOMITANT MEDICATION Use of nonsteroidal anti-inflammatory drug (NSAID), aminoglycocide, cyclosporin, cysplatin will not be allowed within 48 hours prior to PCI and throughout the study duration. Metformin should be withheld 48 hours before and 48 hours after PCI. ACE inhibitors can be continued at the discretion of the doctor in charge. Concomitant medications or treatments received during the study must be reported on the concomitant medication case report form provided.

Study End Points and Statistical Analysis

The primary outcome measure is development of CIN, defined as an increase in serum creatinine of 25% or more within 48 hours after PCI (the efficacy parameter). Post-contrast creatinine will be assessed the mornings of days 1 and 2. The highest serum creatinine on post-contrast days 1 or 2 will be used to calculate the change in serum creatinine.

Trial Size Based on our own and other previous data1,2,4, we assumed the development of CIN of 15% in NAC, 15 % in SOB and 5 % in COM. A group sample size of 210 patients would be required to detect a statistically significant difference with a power of 90% and two-tailed test size of 5% between COM and either of SOB or NAC; giving a total of 630 patients

Final Analysis Analysis will be by intention-to-treat. For the efficacy parameter, a comparison will be made between COM and the average of SOB and NAC (the primary analysis). Pair-wise comparisons may also be made between COM and each of SOB and NAC. Tests for significance will be conducted using the chi-squared test for the primary endpoint. Relative risks and their 95% confidence intervals will be presented for the primary analysis and, although not powered to demonstrate equivalence, between SOB and NAC. Further analysis will be conducted using logistic regression to adjust for potential risk factors. For binary saftey outcomes (need for hemodialysis within 30 days and 30-day mortality) and adverse events, the chi-squared test or Fisher's exact test will be used. T-tests or Wilcoxon-signed rank tests will be used for continuous saftey outcomes (maximum change in serum creatinine level within 30 days, length of hospital stay, maximum change in GFR within 30 days and peak creatinine level within 48 hours and 30 days). A two-tailed significance level of p<0.05 will be used for all endpoints at the final analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 21 year
* Glomerular Filtration Rate (GFR) 15-60ml/min calculated by MDRD formula
* Scheduled to undergo elective PCI
* Able to receive 12 hours of pre-hydration
* Written informed consent

Exclusion Criteria:

* GFR less than 15ml/min or patients diagnosed with end stage renal failure
* Increase in serum creatinine levels of > 0.5mg/dl or 44umol/l in the previous 24 hours
* Preexisting dialysis
* Pulmonary edema or moderate to severe congestive heart failure (New York Heart
* Association [NYHA] III-IV)
* Patient unable to withstand the fluid load and hemodynamics compromise
* Uncontrolled hypertension (untreated systolic blood pressure > 160 mmHg, or diastolic blood pressure > 100mmHg.)
* Emergency cardiac catheterization (i.e. patient presenting with ST segment elevation myocardial infarction undergoing primary angioplasty)
* Recent exposure to radiographic contrast (within two days of the study).
* Allergic to radio-contrast
* Administration of sodium bicarbonate solution or NAC within 48 hours before the PCI.
* Patient unable to give consent
* Clinically vulnerable condition requiring continuous fluid therapy e.g. severe sepsis
* Use of NSAID, aminoglycocide, cyclosporin, cysplatin within 48 hours prior to PCI and throughout the study duration

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 477 (Actual)
Dates: Start 2007-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Development of contrast induced nephropathy (defined as >25% rise in baseline creatinine 48 hours post coronary intervention) | 48 hours

SECONDARY OUTCOMES:
• Maximum change in serum creatinine level • Difference in hospital stay between groups • Need for hemodialysis • mortality • Maximum change in GFR • Peak creatinine level | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Huay C Tan, FAMS FSCAI, Principal Investigator — The Heart Institute, National University Hospital of Singapore
Locations (1):
- The Heart Institute, Singapore, Singapore

REFERENCES:
- [Derived] Chong E, Poh KK, Lu Q, Zhang JJ, Tan N, Hou XM, Ong HY, Azan A, Chen SL, Chen JY, Ali RM, Fang WY, Lau TW, Tan HC. Comparison of combination therapy of high-dose oral N-acetylcysteine and intravenous sodium bicarbonate hydration with individual therapies in the reduction of Contrast-induced Nephropathy during Cardiac Catheterisation and Percutaneous Coronary Intervention (CONTRAST): A multi-centre, randomised, controlled trial. Int J Cardiol. 2015 Dec 15;201:237-42. doi: 10.1016/j.ijcard.2015.07.108. Epub 2015 Aug 5. PMID 26301645